CLINICAL TRIAL: NCT07296978
Title: Delicious, Integrative, Good Nutrition and Fulfillment in Elderly Diet (DIGNIFIED) Programme
Brief Title: Elderly Consumer Survey
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Technology (Other)
Responsible Party: Principal Investigator, Verena Tan Ming Hui, Associate Professor, Singapore Institute of Technology
Other Study IDs: RECAS-0497
Record Dates: First submitted 2025-11-16; First posted 2025-12-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Eating Habits; Food choices; Food preference; Elderly
MeSH Terms: conditions — Feeding Behavior; Food Preferences

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a cross-sectional study, aiming to recruit 200 community-dwelling elderly, aged 60 years and above. Recruitments will be made from St. Luke's ElderCare's (SLEC) active aging hubs around Singapore. The investigators will recruit approximately 70% Chinese, 20% Malay and 10% Indian older adults, that is ethnically-representative of the Singapore population. Interviews will be conducted in-person by the study team's research dietitian, SLEC's nutritionist and dietitians. Responses from elderly subjects will be collected electronically using tablets/laptops.

ELIGIBILITY:
Inclusion Criteria:

- Age 60 years and above

Exclusion Criteria:

* Inability to provide informed consent
* Cognitive impairment (i.e. Alzheimer's disease, dementia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults from St Luke's ElderCare active aging centers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Food habits, dietary practices and preference | Single time point, upon recruitment
  A questionnaire consisting of questions relating to food habits, dietary practices and food preferences will be administered

CONTACTS AND LOCATIONS:
Locations (1):
- St Luke's ElderCare, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plans to make IPD